CLINICAL TRIAL: NCT02230696
Title: Comparative Safety and Efficacy of Two Steroid Treatments in the Relief of the Symptoms of Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Padagis LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRG-NY-14-018
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Results first posted 2021-03-15 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — azelastine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test Product (Experimental): Azelastine Hydrochloride/Fluticasone Propionate Nasal Spray - Perrigo
  Interventions: Drug: Azelastine Hydrochloride/Fluticasone Propionate Nasal Spray
- Reference Product (Active Comparator): Azelastine Hydrochloride/Fluticasone Propionate Nasal Spray - Meda
  Interventions: Drug: Azelastine Hydrochloride/Fluticasone Propionate Nasal Spray
- Placebo Product (Placebo Comparator): Placebo nasal spray
  Interventions: Drug: Placebo nasal spray

INTERVENTIONS:
Drug: Azelastine Hydrochloride/Fluticasone Propionate Nasal Spray — 137 micro-grams Azelastine Hydrochloride, 50 micro-grams Fluticasone Propionate
  Other Names: Perrigo Product
  Arms: Test Product
Drug: Azelastine Hydrochloride/Fluticasone Propionate Nasal Spray — 137 micro-grams Azelastine Hydrochloride, 50 micro-grams Fluticasone Propionate
  Other Names: Reference Listed Drug Product
  Arms: Reference Product
Drug: Placebo nasal spray — Placebo nasal spray
  Arms: Placebo Product

SUMMARY:
To compare safety and efficacy of Perrigo's steroid drug product compared with an FDA approved steroid drug product in the treatment of subjects with seasonal allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

1. Complete the informed consent/assent process.
2. Male or female between 12 to 65 years of age, inclusive.
3. Females of childbearing potential willing to use an acceptable form of birth control during the study.
4. Moderate-to-severe allergic rhinitis.
5. At Visits 1 and 2 have instantaneous and reflective symptom scores sufficient enough to qualify for continued participation in the study
6. Subject must have a history (for 2 or more seasons) of seasonal allergy to at least one allergen known to be present during the study season.
7. Subject must be in general good health with no clinically significant disease or medical procedure other than allergic rhinitis within various time periods prior to Visit 1.
8. Subject must be willing and able to understand and comply with the requirements of the study

Exclusion Criteria:

1. Female who is pregnant or nursing, who is not using or does not agree to use an acceptable form of contraception during the study, or who intends to become pregnant during the study.
2. Subject has a history of hypersensitivity or allergy to any ingredient in the drug products.
3. Subject has any condition or abnormality of the upper airway that, in the opinion of the Investigator, could interfere with administration of the product, evaluation of the subject's condition, or other aspect of the trial.
4. The presence of any nasal mucosal crusting, erosion, ulceration, nasal septum perforation, or any kind of blockage of the nasal passages at screening or randomization.
5. Subject has asthma or a history of asthma requiring chronic treatment within two years of Visit 1.
6. Treatment for oral Candidiasis within 30 days of starting the study, or a current oral Candidiasis infection.
7. Subject has had recent exposure (30 days) or is at risk of being exposed to chicken pox or measles.
8. Subjects with any untreated fungal, bacterial, systemic viral infections within the previous 30 days.
9. Use of various therapies within the given time period prior to Visit 1 and throughout the study.
10. Initiation of hormone replacement therapy during the study.
11. Initiation of immunotherapy during the study, or changes in dosage or frequency of immunotherapy within the 30 days preceding Visit 1.
12. Subject has received immune-system therapy or peptide immunotherapy of any form.
13. Subject had desensitization therapy to the seasonal allergen that is causing their allergic rhinitis within the previous 6 months.
14. Subject presented with conjunctivitis or any other eye signs/symptoms that are not related to the diagnosis of SAR.
15. Clinically relevant abnormal physical findings or medication use within 1 week of randomization, which, in the opinion of the investigator, might interfere with the conduct or results of the study or place the prospective subject at increased risk.
16. Subjects being treated with a product containing a sympathomimetic agent.
17. Subject has previously enrolled in this study or is enrolled in this study with another participating investigator site.
18. Subject is concurrently participating in another investigational study or using any investigational drug (or biologic) or device.
19. Subject plans or anticipates travel outside the local allergen area at any point in the study.
20. History of unresponsiveness to steroid nasal sprays for SAR symptoms.
21. Employee (or employee's family member) of the research center or private practice.
22. If the subject has a smoking history of greater than 10 pack years or has recently started or re-started smoking within the past 2 years

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 951 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Atlanta Allergy & Asthma Clinic, PA, Stockbridge, Georgia
  - Clinical Research Atlanta (CRA), Stockbridge, Georgia
  - Family Allergy and Asthma Research Institute, Louisville, Kentucky
  - Chesapeake Clinical Research, Inc., Baltimore, Maryland
  - NEMRA Northeast Medical Research Associates, Inc, North Dartmouth, Massachusetts
  - Clinical Research Institute, Inc., Minneapolis, Minnesota
  - Clinical Research Institute LLC, Minneapolis, Minnesota
  - Clinical Research of the Ozarks, Inc., Columbia, Missouri
  - Clinical Research of the Ozarks, Inc., Rolla, Missouri
  - The Clinical Research Center, LLC, St Louis, Missouri
  - Princeton Center for Clinical Research, Skillman, New Jersey
  - Island Medical Research, P.C., Rockville Centre, New York
  - Allergy and Asthma Center of NC, High Point, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Toledo Center for Clinical Research, Sylvania, Ohio
  - Allergy, Asthma & Clinical Research Center, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - National Allergy, Asthma & Urticaria Centers of Charleston, North Charleston, South Carolina
  - New Phase Research and Development, Knoxville, Tennessee
  - ISIS Clinical Research, LLC, Austin, Texas
  - Sirius Clinical Research LLC, Austin, Texas
  - AARA Research Center, Dallas, Texas
  - Pharmaceutical Research & Consulting Inc., Dallas, Texas
  - Western Sky Medical Research, El Paso, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Quality Research Inc., San Antonio, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Allergy Asthma Research Institute, Waco, Texas
  - The Asthma & Allergy Center - Bellevue, Bellevue, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Reference Product: Azelastine Hydrochloride/Fluticasone Propionate Nasal Spray Meda
Period: Overall Study
Arm/Group | Test Product | Reference Product | Placebo Product
Started | 381 | 376 | 194
Completed | 366 | 365 | 190
Not Completed | 15 | 11 | 4

BASELINE CHARACTERISTICS:
Groups:
- Test Product: Azelastine Hydrochloride/Fluticasone Propionate Nasal Spray
  Azelastine Hydrochloride/Fluticasone Propionate Nasal Spray: 137 micro-grams Azelastine Hydrochloride, 50 micro-grams Fluticasone Propionate
- Total: Total of all reporting groups
Arm/Group | Test Product | Reference Product | Placebo Product | Total
Number analyzed (Participants) | 381 | 376 | 194 | 951
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (12.87) | 38.6 (13.28) | 38.4 (13.07) | 38.1 (13.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 250 | 248 | 123 | 621
  Male | 131 | 128 | 71 | 330
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52 | 59 | 30 | 141
  Not Hispanic or Latino | 329 | 316 | 164 | 809
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 2 | 7
  Asian | 2 | 2 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 85 | 81 | 41 | 207
  White | 283 | 285 | 148 | 716
  More than one race | 4 | 1 | 0 | 5
  Unknown or Not Reported | 6 | 3 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline for Mean Reflective Total Nasal Symptom Score (rTNSS)
Description: The symptoms included in the reflective Total Nasal Symptom Score (rTNSS) scale are nasal congestion/stuffy nose, nasal discharge/runny nose, sneezing, and itchy nose. Symptoms were scored on a four point scale, 0-3, for each assessment were calculated by totaling these four symptom scores for a maximum score of 12.
Time Frame: Day 1 through Day 14
Population: Per protocol population
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Test Product | Reference Product | Placebo Nasal Spray
Number analyzed (Participants) | 349 | 349 | 181
score on a scale | -2.95 (.15) | -3.13 (.15) | -1.98 (.19)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Equivalence — provides 85% power of success; Trial and Error approach; Equivalence ratio = 94.19, 90% CI 2-sided [84.77 to 104.52]

2. Secondary Outcome: Mean Change From Baseline in the Mean Instantaneous Total Nasal Symptom Score (iTNSS)
Description: The symptoms included in the instantaneous Total Nasal Symptom Score (iTNSS) scale are nasal congestion/stuffy nose, nasal discharge/runny nose, sneezing, and itchy nose. Symptoms were scored on a four point scale, 0-3, for each assessment were calculated by totaling these four symptom scores for a maximum score of 12.
Time Frame: Day 1 through Day 14
Population: per-protocol population
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Test Product | Reference Product | Placebo Nasal Spray
Number analyzed (Participants) | 349 | 349 | 181
score on a scale | -2.81 (0.15) | -2.96 (0.15) | -1.88 (.19)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Equivalence — provides 85% power of success; Trial and Error approach; Equivalence ratio = 94.68, 90% CI 2-sided [84.86 to 105.54]

3. Secondary Outcome: Change From Baseline iTNSS Scores on Day 1 Post First Randomized Dose
Description: This outcome measured the time to statistical significance of the reduction of signs/symptoms over a 4 hour period on Day 1 only by measuring the reduction in iTNSS scores. When the change from baseline was statistically significant, it was associated with a time to onset of the anti-histamine component of the formulation.
  Subjects will record iTNSS scores for 4 hours post first randomized dose. The symptoms included in the instantaneous Total Nasal Symptom Score (iTNSS) scale are nasal congestion/stuffy nose, nasal discharge/runny nose, sneezing, and itchy nose. Symptoms were scored on a four point scale, 0-3, for each assessment were calculated by totaling these four symptom scores for a maximum score of 12.
Time Frame: Day 1, up to four hours post the first dose
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Test Product | Reference Product | Placebo Nasal Spray
Number analyzed (Participants) | 343 | 343 | 181
units on a scale | -3.41 (0.15) | -3.29 (0.15) | -2.94 (.20)

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Test Product | Reference Product | Placebo Product
All-Cause Mortality (participants affected / at risk) | 0/381 | 0/376 | 0/194
Serious Adverse Events (participants affected / at risk) | 3/381 | 1/376 | 0/194
Other Adverse Events (participants affected / at risk) | 0/381 | 0/376 | 0/194
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product (N=381) | Reference Product (N=376) | Placebo Product (N=194)
Fetal demise (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
cervical disc herniation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Infected cat bite (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
suicidal ideations (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2014-09-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT02230696/Prot_001.pdf
  • Statistical Analysis Plan (2014-09-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT02230696/SAP_000.pdf